CLINICAL TRIAL: NCT00005182
Title: Health Professionals Follow-up Study
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Eric B. Rimm, Associate Professor, Harvard School of Public Health (HSPH)
Other Study IDs: 1060; R00HL088372 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Cardiovascular Diseases; Cerebrovascular Accident; Coronary Disease; Peripheral Vascular Diseases; Heart Diseases; Myocardial Infarction
MeSH Terms: conditions — Cardiovascular Diseases; Stroke; Coronary Disease; Peripheral Vascular Diseases; Heart Diseases; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, RBC, WBC

SUMMARY:
To test the hypothesis that increased risk of coronary heart disease, stroke, peripheral vascular disease, and cancer is related to diets high in saturated fat, animal protein, and hydrogenated vegetable oil, and low in polyunsaturated fat, fiber, vitamins A, C, and E, calcium, selenium, and chromium.

DETAILED DESCRIPTION:
BACKGROUND:

The diet-heart hypothesis, that high dietary saturated fat and cholesterol intake increase the risk and high polyunsaturated fat reduces the risk of coronary heart disease in man is supported by ecologic studies, by experiments in rodents and non-human primates, by voluminous literature relating dietary factors to serum lipids, by several secondary prevention trials, and by the Lipid Research Clinics Trial demonstrating a reduction in coronary heart disease among participants assigned to cholestyramine.

Despite the substantial scientific interest and the obvious public health implications of the diet and heart disease issue, relatively few observational cohort or case-control investigations had been published prior to 1985. Although these observational studies were not entirely consistent, taken collectively, they tended to provide important general support for the diet-heart hypothesis. However, due to study design, limited numbers of endpoints, or methods of analysis, many central questions remained unanswered. The most important issue was the quantitative relationship between specific dietary factors and risk of coronary heart disease. Moreover, the interplay of dietary and genetic factors is poorly understood.

DESIGN NARRATIVE:

In this prospective cohort study, participants completed a mailed general medical and health questionnaire at baseline and an intensively validated semiquantitative food frequency questionnaire (SFFQ). At one year, tissue specimens were collected and catalogued for future nested case-control analyses of coronary heart disease risk in relation to levels of calcium, selenium, and chromium. Follow-up questionnaires to update exposure information and ascertain non-fatal endpoints were mailed at two-year intervals. All reported cases of non-fatal myocardial infarction, stroke, and cancer were documented with hospital records and/or pathology reports. Fatal events were ascertained with the National Death Index and documented. To standardize SFFQ nutrient scores against measurements of absolute intake, two one-week diet records were obtained from a random sample of 150 Boston-area participants.

The study was renewed in 1991, 1997, and in 2003 to continue the follow-up of 51,529 male health professionals. The cohort is followed by questionnaires mailed at two-year intervals to update exposure information and ascertain nonfatal events. Complete dietary assessments are included every four years.A subset of 18,225 participants provided blood samples between 1993 and 1995. Genotyping was performed among 435 cardiovascular disease cases and 878 controls using Affymetrix 6.0 platform.

ELIGIBILITY:
Recruited through their professional organizations or occupation from mailing house lists.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male Health Professionals
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 1985-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Incident CVD | Renewed every 5 years since 1986

CONTACTS AND LOCATIONS:
Overall Officials: Eric Rimm, Principal Investigator — Harvard School of Public Health (HSPH)

REFERENCES:
- [Background] MacIntosh DL, Williams PL, Hunter DJ, Sampson LA, Morris SC, Willett WC, Rimm EB. Evaluation of a food frequency questionnaire-food composition approach for estimating dietary intake of inorganic arsenic and methylmercury. Cancer Epidemiol Biomarkers Prev. 1997 Dec;6(12):1043-50. PMID 9419401
- [Background] Giovannucci E, Rimm EB, Wolk A, Ascherio A, Stampfer MJ, Colditz GA, Willett WC. Calcium and fructose intake in relation to risk of prostate cancer. Cancer Res. 1998 Feb 1;58(3):442-7. PMID 9458087
- [Background] Welch G, Kawachi I, Barry MJ, Giovannucci E, Colditz GA, Willett WC. Distinction between symptoms of voiding and filling in benign prostatic hyperplasia: findings from the Health Professionals Follow-up Study. Urology. 1998 Mar;51(3):422-7. doi: 10.1016/s0090-4295(97)00626-2. PMID 9510347
- [Background] Madore F, Stampfer MJ, Rimm EB, Curhan GC. Nephrolithiasis and risk of hypertension. Am J Hypertens. 1998 Jan;11(1 Pt 1):46-53. doi: 10.1016/s0895-7061(97)00371-3. PMID 9504449
- [Background] Giovannucci E, Rimm EB, Stampfer MJ, Colditz GA, Willett WC. Diabetes mellitus and risk of prostate cancer (United States). Cancer Causes Control. 1998 Jan;9(1):3-9. doi: 10.1023/a:1008822917449. PMID 9486458
- [Background] Coakley EH, Rimm EB, Colditz G, Kawachi I, Willett W. Predictors of weight change in men: results from the Health Professionals Follow-up Study. Int J Obes Relat Metab Disord. 1998 Feb;22(2):89-96. doi: 10.1038/sj.ijo.0800549. PMID 9504316
- [Background] Aldoori WH, Giovannucci EL, Rockett HR, Sampson L, Rimm EB, Willett WC. A prospective study of dietary fiber types and symptomatic diverticular disease in men. J Nutr. 1998 Apr;128(4):714-9. doi: 10.1093/jn/128.4.714. PMID 9521633
- [Background] Aldoori WH, Giovannucci EL, Rimm EB, Wing AL, Willett WC. Use of acetaminophen and nonsteroidal anti-inflammatory drugs: a prospective study and the risk of symptomatic diverticular disease in men. Arch Fam Med. 1998 May-Jun;7(3):255-60. doi: 10.1001/archfami.7.3.255. PMID 9596460
- [Background] Rosner B, Willett WC. Interval estimates for correlation coefficients corrected for within-person variation: implications for study design and hypothesis testing. Am J Epidemiol. 1988 Feb;127(2):377-86. doi: 10.1093/oxfordjournals.aje.a114811. PMID 3337089
- [Background] Rimm EB, Stampfer MJ, Colditz GA, Giovannucci E, Willett WC. Effectiveness of various mailing strategies among nonrespondents in a prospective cohort study. Am J Epidemiol. 1990 Jun;131(6):1068-71. doi: 10.1093/oxfordjournals.aje.a115598. PMID 2343859
- [Background] Hunter DJ, Rimm EB, Sacks FM, Stampfer MJ, Colditz GA, Litin LB, Willett WC. Comparison of measures of fatty acid intake by subcutaneous fat aspirate, food frequency questionnaire, and diet records in a free-living population of US men. Am J Epidemiol. 1992 Feb 15;135(4):418-27. doi: 10.1093/oxfordjournals.aje.a116302. PMID 1550093
- [Background] Rimm EB, Giovannucci EL, Willett WC, Colditz GA, Ascherio A, Rosner B, Stampfer MJ. Prospective study of alcohol consumption and risk of coronary disease in men. Lancet. 1991 Aug 24;338(8765):464-8. doi: 10.1016/0140-6736(91)90542-w. PMID 1678444
- [Background] Ascherio A, Stampfer MJ, Colditz GA, Willett WC, McKinlay J. Nutrient intakes and blood pressure in normotensive males. Int J Epidemiol. 1991 Dec;20(4):886-91. doi: 10.1093/ije/20.4.886. PMID 1666065
- [Background] Giovannucci E, Colditz G, Stampfer MJ, Rimm EB, Litin L, Sampson L, Willett WC. The assessment of alcohol consumption by a simple self-administered questionnaire. Am J Epidemiol. 1991 Apr 15;133(8):810-7. doi: 10.1093/oxfordjournals.aje.a115960. PMID 2021148
- [Background] Colditz GA, Rimm EB, Giovannucci E, Stampfer MJ, Rosner B, Willett WC. A prospective study of parental history of myocardial infarction and coronary artery disease in men. Am J Cardiol. 1991 May 1;67(11):933-8. doi: 10.1016/0002-9149(91)90163-f. PMID 2018010
- [Background] Ching PL, Willett WC, Rimm EB, Colditz GA, Gortmaker SL, Stampfer MJ. Activity level and risk of overweight in male health professionals. Am J Public Health. 1996 Jan;86(1):25-30. doi: 10.2105/ajph.86.1.25. PMID 8561237
- [Background] Curhan GC, Willett WC, Rimm EB, Spiegelman D, Stampfer MJ. Prospective study of beverage use and the risk of kidney stones. Am J Epidemiol. 1996 Feb 1;143(3):240-7. doi: 10.1093/oxfordjournals.aje.a008734. PMID 8561157
- [Background] Giovannucci E, Ascherio A, Rimm EB, Stampfer MJ, Colditz GA, Willett WC. Intake of carotenoids and retinol in relation to risk of prostate cancer. J Natl Cancer Inst. 1995 Dec 6;87(23):1767-76. doi: 10.1093/jnci/87.23.1767. PMID 7473833
- [Background] Giovannucci E, Rimm EB, Chute CG, Kawachi I, Colditz GA, Stampfer MJ, Willett WC. Obesity and benign prostatic hyperplasia. Am J Epidemiol. 1994 Dec 1;140(11):989-1002. doi: 10.1093/oxfordjournals.aje.a117206. PMID 7527182
- [Background] Aldoori WH, Giovannucci EL, Rimm EB, Wing AL, Trichopoulos DV, Willett WC. A prospective study of alcohol, smoking, caffeine, and the risk of symptomatic diverticular disease in men. Ann Epidemiol. 1995 May;5(3):221-8. doi: 10.1016/1047-2797(94)00109-7. PMID 7606311
- [Background] Rimm EB, Stampfer MJ, Giovannucci E, Ascherio A, Spiegelman D, Colditz GA, Willett WC. Body size and fat distribution as predictors of coronary heart disease among middle-aged and older US men. Am J Epidemiol. 1995 Jun 15;141(12):1117-27. doi: 10.1093/oxfordjournals.aje.a117385. PMID 7771450
- [Background] Kearney J, Giovannucci E, Rimm EB, Stampfer MJ, Colditz GA, Ascherio A, Bleday R, Willett WC. Diet, alcohol, and smoking and the occurrence of hyperplastic polyps of the colon and rectum (United States). Cancer Causes Control. 1995 Jan;6(1):45-56. doi: 10.1007/BF00051680. PMID 7718735
- [Background] Giovannucci E, Rimm EB, Ascherio A, Stampfer MJ, Colditz GA, Willett WC. Alcohol, low-methionine--low-folate diets, and risk of colon cancer in men. J Natl Cancer Inst. 1995 Feb 15;87(4):265-73. doi: 10.1093/jnci/87.4.265. PMID 7707417
- [Background] Rimm EB, Chan J, Stampfer MJ, Colditz GA, Willett WC. Prospective study of cigarette smoking, alcohol use, and the risk of diabetes in men. BMJ. 1995 Mar 4;310(6979):555-9. doi: 10.1136/bmj.310.6979.555. PMID 7888928
- [Background] Ascherio A, Rimm EB, Stampfer MJ, Giovannucci EL, Willett WC. Dietary intake of marine n-3 fatty acids, fish intake, and the risk of coronary disease among men. N Engl J Med. 1995 Apr 13;332(15):977-82. doi: 10.1056/NEJM199504133321501. PMID 7885425
- [Background] Aldoori WH, Giovannucci EL, Rimm EB, Ascherio A, Stampfer MJ, Colditz GA, Wing AL, Trichopoulos DV, Willett WC. Prospective study of physical activity and the risk of symptomatic diverticular disease in men. Gut. 1995 Feb;36(2):276-82. doi: 10.1136/gut.36.2.276. PMID 7883230
- [Background] Giovannucci E, Ascherio A, Rimm EB, Colditz GA, Stampfer MJ, Willett WC. Physical activity, obesity, and risk for colon cancer and adenoma in men. Ann Intern Med. 1995 Mar 1;122(5):327-34. doi: 10.7326/0003-4819-122-5-199503010-00002. PMID 7847643
- [Background] Chan JM, Rimm EB, Colditz GA, Stampfer MJ, Willett WC. Obesity, fat distribution, and weight gain as risk factors for clinical diabetes in men. Diabetes Care. 1994 Sep;17(9):961-9. doi: 10.2337/diacare.17.9.961. PMID 7988316
- [Background] Aldoori WH, Giovannucci EL, Rimm EB, Wing AL, Trichopoulos DV, Willett WC. A prospective study of diet and the risk of symptomatic diverticular disease in men. Am J Clin Nutr. 1994 Nov;60(5):757-64. doi: 10.1093/ajcn/60.5.757. PMID 7942584
- [Background] Hemenway D, Azrael DR, Rimm EB, Feskanich D, Willett WC. Risk factors for wrist fracture: effect of age, cigarettes, alcohol, body height, relative weight, and handedness on the risk for distal forearm fractures in men. Am J Epidemiol. 1994 Aug 15;140(4):361-7. doi: 10.1093/oxfordjournals.aje.a117258. PMID 8059771
- [Background] Giovannucci E, Rimm EB, Stampfer MJ, Colditz GA, Ascherio A, Willett WC. Aspirin use and the risk for colorectal cancer and adenoma in male health professionals. Ann Intern Med. 1994 Aug 15;121(4):241-6. doi: 10.7326/0003-4819-121-4-199408150-00001. PMID 8037405
- [Background] Kawachi I, Colditz GA, Ascherio A, Rimm EB, Giovannucci E, Stampfer MJ, Willett WC. Prospective study of phobic anxiety and risk of coronary heart disease in men. Circulation. 1994 May;89(5):1992-7. doi: 10.1161/01.cir.89.5.1992. PMID 8181122
- [Background] Giovannucci E, Rimm EB, Stampfer MJ, Colditz GA, Ascherio A, Willett WC. Intake of fat, meat, and fiber in relation to risk of colon cancer in men. Cancer Res. 1994 May 1;54(9):2390-7. PMID 8162586
- [Background] Curhan GC, Rimm EB, Willett WC, Stampfer MJ. Regional variation in nephrolithiasis incidence and prevalence among United States men. J Urol. 1994 Apr;151(4):838-41. doi: 10.1016/s0022-5347(17)35101-7. PMID 8126805
- [Background] Ascherio A, Willett WC, Rimm EB, Giovannucci EL, Stampfer MJ. Dietary iron intake and risk of coronary disease among men. Circulation. 1994 Mar;89(3):969-74. doi: 10.1161/01.cir.89.3.969. PMID 8124837
- [Background] Giovannucci E, Rimm EB, Stampfer MJ, Colditz GA, Ascherio A, Kearney J, Willett WC. A prospective study of cigarette smoking and risk of colorectal adenoma and colorectal cancer in U.S. men. J Natl Cancer Inst. 1994 Feb 2;86(3):183-91. doi: 10.1093/jnci/86.3.183. PMID 8283490
- [Background] Feskanich D, Rimm EB, Giovannucci EL, Colditz GA, Stampfer MJ, Litin LB, Willett WC. Reproducibility and validity of food intake measurements from a semiquantitative food frequency questionnaire. J Am Diet Assoc. 1993 Jul;93(7):790-6. doi: 10.1016/0002-8223(93)91754-e. PMID 8320406
- [Background] Rimm E, Colditz G. Smoking, alcohol, and plasma levels of carotenes and vitamin E. Ann N Y Acad Sci. 1993 May 28;686:323-33; discussion 333-4. doi: 10.1111/j.1749-6632.1993.tb39195.x. PMID 8512258
- [Background] Rimm EB, Stampfer MJ, Ascherio A, Giovannucci E, Colditz GA, Willett WC. Vitamin E consumption and the risk of coronary heart disease in men. N Engl J Med. 1993 May 20;328(20):1450-6. doi: 10.1056/NEJM199305203282004. PMID 8479464
- [Background] Curhan GC, Willett WC, Rimm EB, Stampfer MJ. A prospective study of dietary calcium and other nutrients and the risk of symptomatic kidney stones. N Engl J Med. 1993 Mar 25;328(12):833-8. doi: 10.1056/NEJM199303253281203. PMID 8441427
- [Background] Giovannucci E, Ascherio A, Rimm EB, Colditz GA, Stampfer MJ, Willett WC. A prospective cohort study of vasectomy and prostate cancer in US men. JAMA. 1993 Feb 17;269(7):873-7. PMID 8426446
- [Background] Kearney J, Giovannucci E, Rimm EB, Ascherio A, Stampfer MJ, Colditz GA, Wing A, Kampman E, Willett WC. Calcium, vitamin D, and dairy foods and the occurrence of colon cancer in men. Am J Epidemiol. 1996 May 1;143(9):907-17. doi: 10.1093/oxfordjournals.aje.a008834. PMID 8610704
- [Background] Stampfer MJ, Rimm EB. Folate and cardiovascular disease. Why we need a trial now. JAMA. 1996 Jun 26;275(24):1929-30. No abstract available. PMID 8648876
- [Background] Chasan-Taber S, Rimm EB, Stampfer MJ, Spiegelman D, Colditz GA, Giovannucci E, Ascherio A, Willett WC. Reproducibility and validity of a self-administered physical activity questionnaire for male health professionals. Epidemiology. 1996 Jan;7(1):81-6. doi: 10.1097/00001648-199601000-00014. PMID 8664406
- [Background] Willett WC. Diet, nutrition, and avoidable cancer. Environ Health Perspect. 1995 Nov;103 Suppl 8(Suppl 8):165-70. doi: 10.1289/ehp.95103s8165. PMID 8741778
- [Background] Joshipura KJ, Willett WC, Douglass CW. The impact of edentulousness on food and nutrient intake. J Am Dent Assoc. 1996 Apr;127(4):459-67. doi: 10.14219/jada.archive.1996.0237. PMID 8655866
- [Background] Curhan GC, Willett WC, Rimm EB, Stampfer MJ. A prospective study of the intake of vitamins C and B6, and the risk of kidney stones in men. J Urol. 1996 Jun;155(6):1847-51. PMID 8618271
- [Background] Rimm EB, Ascherio A, Giovannucci E, Spiegelman D, Stampfer MJ, Willett WC. Vegetable, fruit, and cereal fiber intake and risk of coronary heart disease among men. JAMA. 1996 Feb 14;275(6):447-51. doi: 10.1001/jama.1996.03530300031036. PMID 8627965
- [Background] Ascherio A, Rimm EB, Giovannucci EL, Spiegelman D, Stampfer M, Willett WC. Dietary fat and risk of coronary heart disease in men: cohort follow up study in the United States. BMJ. 1996 Jul 13;313(7049):84-90. doi: 10.1136/bmj.313.7049.84. PMID 8688759
- [Background] Joshipura KJ, Rimm EB, Douglass CW, Trichopoulos D, Ascherio A, Willett WC. Poor oral health and coronary heart disease. J Dent Res. 1996 Sep;75(9):1631-6. doi: 10.1177/00220345960750090301. PMID 8952614
- [Background] Walker SP, Rimm EB, Ascherio A, Kawachi I, Stampfer MJ, Willett WC. Body size and fat distribution as predictors of stroke among US men. Am J Epidemiol. 1996 Dec 15;144(12):1143-50. doi: 10.1093/oxfordjournals.aje.a008892. PMID 8956626
- [Background] Aldoori WH, Giovannucci EL, Stampfer MJ, Rimm EB, Wing AL, Willett WC. Prospective study of diet and the risk of duodenal ulcer in men. Am J Epidemiol. 1997 Jan 1;145(1):42-50. doi: 10.1093/oxfordjournals.aje.a009030. PMID 8982021
- [Background] Curhan GC, Willett WC, Rimm EB, Spiegelman D, Ascherio AL, Stampfer MJ. Birth weight and adult hypertension, diabetes mellitus, and obesity in US men. Circulation. 1996 Dec 15;94(12):3246-50. doi: 10.1161/01.cir.94.12.3246. PMID 8989136
- [Background] Joshipura KJ, Douglass CW, Garcia RI, Valachovic R, Willett WC. Validity of a self-reported periodontal disease measure. J Public Health Dent. 1996 Summer;56(4):205-12. doi: 10.1111/j.1752-7325.1996.tb02437.x. PMID 8906704
- [Background] Kawachi I, Barry MJ, Giovannucci E, Rimm EB, Colditz GA, Stampfer MJ, Willett WC. The impact of different therapies on symptoms of benign prostatic hyperplasia: a prospective study. Clin Ther. 1996 Nov-Dec;18(6):1118-27. doi: 10.1016/s0149-2918(96)80066-x. PMID 9001828
- [Background] Salmeron J, Ascherio A, Rimm EB, Colditz GA, Spiegelman D, Jenkins DJ, Stampfer MJ, Wing AL, Willett WC. Dietary fiber, glycemic load, and risk of NIDDM in men. Diabetes Care. 1997 Apr;20(4):545-50. doi: 10.2337/diacare.20.4.545. PMID 9096978
- [Background] Kawachi I, Colditz GA, Ascherio A, Rimm EB, Giovannucci E, Stampfer MJ, Willett WC. A prospective study of social networks in relation to total mortality and cardiovascular disease in men in the USA. J Epidemiol Community Health. 1996 Jun;50(3):245-51. doi: 10.1136/jech.50.3.245. PMID 8935453
- [Background] Aldoori WH, Giovannucci EL, Stampfer MJ, Rimm EB, Wing AL, Willett WC. A prospective study of alcohol, smoking, caffeine, and the risk of duodenal ulcer in men. Epidemiology. 1997 Jul;8(4):420-4. doi: 10.1097/00001648-199707000-00012. PMID 9209857
- [Background] Platz EA, Giovannucci E, Rimm EB, Rockett HR, Stampfer MJ, Colditz GA, Willett WC. Dietary fiber and distal colorectal adenoma in men. Cancer Epidemiol Biomarkers Prev. 1997 Sep;6(9):661-70. PMID 9298572
- [Background] Owusu W, Willett WC, Feskanich D, Ascherio A, Spiegelman D, Colditz GA. Calcium intake and the incidence of forearm and hip fractures among men. J Nutr. 1997 Sep;127(9):1782-7. doi: 10.1093/jn/127.9.1782. PMID 9278560
- [Background] Curhan GC, Willett WC, Rimm EB, Stampfer MJ. Family history and risk of kidney stones. J Am Soc Nephrol. 1997 Oct;8(10):1568-73. doi: 10.1681/ASN.V8101568. PMID 9335385
- [Background] Miller M, Hemenway D, Rimm E. Cigarettes and suicide: a prospective study of 50,000 men. Am J Public Health. 2000 May;90(5):768-73. doi: 10.2105/ajph.90.5.768. PMID 10800427
- [Background] Platz EA, Kawachi I, Rimm EB, Willett WC, Giovannucci E. Race, ethnicity and benign prostatic hyperplasia in the health professionals follow-up study. J Urol. 2000 Feb;163(2):490-5. PMID 10647663
- [Background] van Dam RM, Huang Z, Giovannucci E, Rimm EB, Hunter DJ, Colditz GA, Stampfer MJ, Willett WC. Diet and basal cell carcinoma of the skin in a prospective cohort of men. Am J Clin Nutr. 2000 Jan;71(1):135-41. doi: 10.1093/ajcn/71.1.135. PMID 10617958
- [Background] Platz EA, Pollak MN, Rimm EB, Majeed N, Tao Y, Willett WC, Giovannucci E. Racial variation in insulin-like growth factor-1 and binding protein-3 concentrations in middle-aged men. Cancer Epidemiol Biomarkers Prev. 1999 Dec;8(12):1107-10. PMID 10613344
- [Background] Brown L, Rimm EB, Seddon JM, Giovannucci EL, Chasan-Taber L, Spiegelman D, Willett WC, Hankinson SE. A prospective study of carotenoid intake and risk of cataract extraction in US men. Am J Clin Nutr. 1999 Oct;70(4):517-24. doi: 10.1093/ajcn/70.4.517. PMID 10500021
- [Background] Meigs JB, Barry MJ, Giovannucci E, Rimm EB, Stampfer MJ, Kawachi I. Incidence rates and risk factors for acute urinary retention: the health professionals followup study. J Urol. 1999 Aug;162(2):376-82. PMID 10411042
- [Background] Ascherio A, Rimm EB, Hernan MA, Giovannucci E, Kawachi I, Stampfer MJ, Willett WC. Relation of consumption of vitamin E, vitamin C, and carotenoids to risk for stroke among men in the United States. Ann Intern Med. 1999 Jun 15;130(12):963-70. doi: 10.7326/0003-4819-130-12-199906150-00003. PMID 10383366
- [Background] Leitzmann MF, Giovannucci EL, Stampfer MJ, Spiegelman D, Colditz GA, Willett WC, Rimm EB. Prospective study of alcohol consumption patterns in relation to symptomatic gallstone disease in men. Alcohol Clin Exp Res. 1999 May;23(5):835-41. PMID 10371403
- [Background] Leitzmann MF, Willett WC, Rimm EB, Stampfer MJ, Spiegelman D, Colditz GA, Giovannucci E. A prospective study of coffee consumption and the risk of symptomatic gallstone disease in men. JAMA. 1999 Jun 9;281(22):2106-12. doi: 10.1001/jama.281.22.2106. PMID 10367821
- [Background] Ascherio A, Rimm EB, Hernan MA, Giovannucci EL, Kawachi I, Stampfer MJ, Willett WC. Intake of potassium, magnesium, calcium, and fiber and risk of stroke among US men. Circulation. 1998 Sep 22;98(12):1198-204. doi: 10.1161/01.cir.98.12.1198. PMID 9743511
- [Background] Curhan GC, Willett WC, Rimm EB, Speizer FE, Stampfer MJ. Body size and risk of kidney stones. J Am Soc Nephrol. 1998 Sep;9(9):1645-52. doi: 10.1681/ASN.V991645. PMID 9727373
- [Background] Verhoef P, Rimm EB, Hunter DJ, Chen J, Willett WC, Kelsey K, Stampfer MJ. A common mutation in the methylenetetrahydrofolate reductase gene and risk of coronary heart disease: results among U.S. men. J Am Coll Cardiol. 1998 Aug;32(2):353-9. doi: 10.1016/s0735-1097(98)00244-7. PMID 9708460
- [Background] Chu NF, Spiegelman D, Rifai N, Hotamisligil GS, Rimm EB. Glycemic status and soluble tumor necrosis factor receptor levels in relation to plasma leptin concentrations among normal weight and overweight US men. Int J Obes Relat Metab Disord. 2000 Sep;24(9):1085-92. doi: 10.1038/sj.ijo.0801361. PMID 11033975
- [Background] Hu FB, Rimm EB, Stampfer MJ, Ascherio A, Spiegelman D, Willett WC. Prospective study of major dietary patterns and risk of coronary heart disease in men. Am J Clin Nutr. 2000 Oct;72(4):912-21. doi: 10.1093/ajcn/72.4.912. PMID 11010931
- [Background] Ascherio A, Rimm EB, Giovannucci E, Willett WC, Stampfer MJ. Blood donations and risk of coronary heart disease in men. Circulation. 2001 Jan 2;103(1):52-7. doi: 10.1161/01.cir.103.1.52. PMID 11136685
- [Background] Fung TT, Hu FB, Yu J, Chu NF, Spiegelman D, Tofler GH, Willett WC, Rimm EB. Leisure-time physical activity, television watching, and plasma biomarkers of obesity and cardiovascular disease risk. Am J Epidemiol. 2000 Dec 15;152(12):1171-8. doi: 10.1093/aje/152.12.1171. PMID 11130623
- [Background] Fung TT, Rimm EB, Spiegelman D, Rifai N, Tofler GH, Willett WC, Hu FB. Association between dietary patterns and plasma biomarkers of obesity and cardiovascular disease risk. Am J Clin Nutr. 2001 Jan;73(1):61-7. doi: 10.1093/ajcn/73.1.61. PMID 11124751
- [Background] McCullough ML, Feskanich D, Rimm EB, Giovannucci EL, Ascherio A, Variyam JN, Spiegelman D, Stampfer MJ, Willett WC. Adherence to the Dietary Guidelines for Americans and risk of major chronic disease in men. Am J Clin Nutr. 2000 Nov;72(5):1223-31. doi: 10.1093/ajcn/72.5.1223. PMID 11063453
- [Background] Joshipura KJ, Ascherio A, Manson JE, Stampfer MJ, Rimm EB, Speizer FE, Hennekens CH, Spiegelman D, Willett WC. Fruit and vegetable intake in relation to risk of ischemic stroke. JAMA. 1999 Oct 6;282(13):1233-9. doi: 10.1001/jama.282.13.1233. PMID 10517425
- [Background] Willett W, Stampfer M, Chu NF, Spiegelman D, Holmes M, Rimm E. Assessment of questionnaire validity for measuring total fat intake using plasma lipid levels as criteria. Am J Epidemiol. 2001 Dec 15;154(12):1107-12. doi: 10.1093/aje/154.12.1107. PMID 11744515
- [Background] Conigrave KM, Hu BF, Camargo CA Jr, Stampfer MJ, Willett WC, Rimm EB. A prospective study of drinking patterns in relation to risk of type 2 diabetes among men. Diabetes. 2001 Oct;50(10):2390-5. doi: 10.2337/diabetes.50.10.2390. PMID 11574424
- [Background] Chu NF, Spiegelman D, Hotamisligil GS, Rifai N, Stampfer M, Rimm EB. Plasma insulin, leptin, and soluble TNF receptors levels in relation to obesity-related atherogenic and thrombogenic cardiovascular disease risk factors among men. Atherosclerosis. 2001 Aug;157(2):495-503. doi: 10.1016/s0021-9150(00)00755-3. PMID 11472752
- [Background] Field AE, Coakley EH, Must A, Spadano JL, Laird N, Dietz WH, Rimm E, Colditz GA. Impact of overweight on the risk of developing common chronic diseases during a 10-year period. Arch Intern Med. 2001 Jul 9;161(13):1581-6. doi: 10.1001/archinte.161.13.1581. PMID 11434789
- [Background] Hu FB, Willett WC. Diet and coronary heart disease: findings from the Nurses' Health Study and Health Professionals' Follow-up Study. J Nutr Health Aging. 2001;5(3):132-8. PMID 11458281
- [Background] Hu FB, Leitzmann MF, Stampfer MJ, Colditz GA, Willett WC, Rimm EB. Physical activity and television watching in relation to risk for type 2 diabetes mellitus in men. Arch Intern Med. 2001 Jun 25;161(12):1542-8. doi: 10.1001/archinte.161.12.1542. PMID 11427103
- [Background] Joshipura KJ, Hu FB, Manson JE, Stampfer MJ, Rimm EB, Speizer FE, Colditz G, Ascherio A, Rosner B, Spiegelman D, Willett WC. The effect of fruit and vegetable intake on risk for coronary heart disease. Ann Intern Med. 2001 Jun 19;134(12):1106-14. doi: 10.7326/0003-4819-134-12-200106190-00010. PMID 11412050
- [Background] Chu NF, Spiegelman D, Yu J, Rifai N, Hotamisligil GS, Rimm EB. Plasma leptin concentrations and four-year weight gain among US men. Int J Obes Relat Metab Disord. 2001 Mar;25(3):346-53. doi: 10.1038/sj.ijo.0801549. PMID 11319631
- [Background] Chu NF, Stampfer MJ, Spiegelman D, Rifai N, Hotamisligil GS, Rimm EB. Dietary and lifestyle factors in relation to plasma leptin concentrations among normal weight and overweight men. Int J Obes Relat Metab Disord. 2001 Jan;25(1):106-14. doi: 10.1038/sj.ijo.0801468. PMID 11244465
- [Background] van Dam RM, Willett WC, Rimm EB, Stampfer MJ, Hu FB. Dietary fat and meat intake in relation to risk of type 2 diabetes in men. Diabetes Care. 2002 Mar;25(3):417-24. doi: 10.2337/diacare.25.3.417. PMID 11874924
- [Background] van Dam RM, Rimm EB, Willett WC, Stampfer MJ, Hu FB. Dietary patterns and risk for type 2 diabetes mellitus in U.S. men. Ann Intern Med. 2002 Feb 5;136(3):201-9. doi: 10.7326/0003-4819-136-3-200202050-00008. PMID 11827496
- [Background] Fung TT, Hu FB, Pereira MA, Liu S, Stampfer MJ, Colditz GA, Willett WC. Whole-grain intake and the risk of type 2 diabetes: a prospective study in men. Am J Clin Nutr. 2002 Sep;76(3):535-40. doi: 10.1093/ajcn/76.3.535. PMID 12197996
- [Background] Eng PM, Rimm EB, Fitzmaurice G, Kawachi I. Social ties and change in social ties in relation to subsequent total and cause-specific mortality and coronary heart disease incidence in men. Am J Epidemiol. 2002 Apr 15;155(8):700-9. doi: 10.1093/aje/155.8.700. PMID 11943687
- [Background] Grobbee DE, Rimm EB, Giovannucci E, Colditz G, Stampfer M, Willett W. Coffee, caffeine, and cardiovascular disease in men. N Engl J Med. 1990 Oct 11;323(15):1026-32. doi: 10.1056/NEJM199010113231504. PMID 2215561
- [Background] Bacon CG, Hu FB, Giovannucci E, Glasser DB, Mittleman MA, Rimm EB. Association of type and duration of diabetes with erectile dysfunction in a large cohort of men. Diabetes Care. 2002 Aug;25(8):1458-63. doi: 10.2337/diacare.25.8.1458. PMID 12145250
- [Background] Cho E, Rimm EB, Stampfer MJ, Willett WC, Hu FB. The impact of diabetes mellitus and prior myocardial infarction on mortality from all causes and from coronary heart disease in men. J Am Coll Cardiol. 2002 Sep 4;40(5):954-60. doi: 10.1016/s0735-1097(02)02044-2. PMID 12225722
- [Background] Tanasescu M, Leitzmann MF, Rimm EB, Willett WC, Stampfer MJ, Hu FB. Exercise type and intensity in relation to coronary heart disease in men. JAMA. 2002 Oct 23-30;288(16):1994-2000. doi: 10.1001/jama.288.16.1994. PMID 12387651
- [Background] He K, Rimm EB, Merchant A, Rosner BA, Stampfer MJ, Willett WC, Ascherio A. Fish consumption and risk of stroke in men. JAMA. 2002 Dec 25;288(24):3130-6. doi: 10.1001/jama.288.24.3130. PMID 12495393
- [Background] Goldberg IJ. To drink or not to drink? N Engl J Med. 2003 Jan 9;348(2):163-4. doi: 10.1056/NEJMe020163. No abstract available. PMID 12519927
- [Background] Yoshizawa K, Rimm EB, Morris JS, Spate VL, Hsieh CC, Spiegelman D, Stampfer MJ, Willett WC. Mercury and the risk of coronary heart disease in men. N Engl J Med. 2002 Nov 28;347(22):1755-60. doi: 10.1056/NEJMoa021437. PMID 12456851
- [Background] Mukamal KJ, Conigrave KM, Mittleman MA, Camargo CA Jr, Stampfer MJ, Willett WC, Rimm EB. Roles of drinking pattern and type of alcohol consumed in coronary heart disease in men. N Engl J Med. 2003 Jan 9;348(2):109-18. doi: 10.1056/NEJMoa022095. PMID 12519921
- [Background] Hung HC, Willett W, Merchant A, Rosner BA, Ascherio A, Joshipura KJ. Oral health and peripheral arterial disease. Circulation. 2003 Mar 4;107(8):1152-7. doi: 10.1161/01.cir.0000051456.68470.c8. PMID 12615794
- [Background] Al-Delaimy WK, Rimm E, Willett WC, Stampfer MJ, Hu FB. A prospective study of calcium intake from diet and supplements and risk of ischemic heart disease among men. Am J Clin Nutr. 2003 Apr;77(4):814-8. doi: 10.1093/ajcn/77.4.814. PMID 12663277
- [Background] Tanasescu M, Leitzmann MF, Rimm EB, Hu FB. Physical activity in relation to cardiovascular disease and total mortality among men with type 2 diabetes. Circulation. 2003 May 20;107(19):2435-9. doi: 10.1161/01.CIR.0000066906.11109.1F. Epub 2003 Apr 28. PMID 12719277
- [Background] Pischon T, Hotamisligil GS, Rimm EB. Adiponectin: stability in plasma over 36 hours and within-person variation over 1 year. Clin Chem. 2003 Apr;49(4):650-2. doi: 10.1373/49.4.650. No abstract available. PMID 12651819
- [Background] Joshi A, Douglass CW, Kim HD, Joshipura KJ, Park MC, Rimm EB, Carino MJ, Garcia RI, Morris JS, Willett WC. The relationship between amalgam restorations and mercury levels in male dentists and nondental health professionals. J Public Health Dent. 2003 Winter;63(1):52-60. doi: 10.1111/j.1752-7325.2003.tb03474.x. PMID 12597586
- [Background] Augustsson K, Michaud DS, Rimm EB, Leitzmann MF, Stampfer MJ, Willett WC, Giovannucci E. A prospective study of intake of fish and marine fatty acids and prostate cancer. Cancer Epidemiol Biomarkers Prev. 2003 Jan;12(1):64-7. PMID 12540506
- [Background] Joshipura KJ, Hung HC, Rimm EB, Willett WC, Ascherio A. Periodontal disease, tooth loss, and incidence of ischemic stroke. Stroke. 2003 Jan;34(1):47-52. doi: 10.1161/01.str.0000052974.79428.0c. PMID 12511749
- [Background] Pischon T, Hankinson SE, Hotamisligil GS, Rifai N, Willett WC, Rimm EB. Habitual dietary intake of n-3 and n-6 fatty acids in relation to inflammatory markers among US men and women. Circulation. 2003 Jul 15;108(2):155-60. doi: 10.1161/01.CIR.0000079224.46084.C2. Epub 2003 Jun 23. PMID 12821543
- [Background] Meyer KA, Conigrave KM, Chu NF, Rifai N, Spiegelman D, Stampfer MJ, Rimm EB. Alcohol consumption patterns and HbA1c, C-peptide and insulin concentrations in men. J Am Coll Nutr. 2003 Jun;22(3):185-94. doi: 10.1080/07315724.2003.10719292. PMID 12805244
- [Background] Yoshizawa K, Ascherio A, Morris JS, Stampfer MJ, Giovannucci E, Baskett CK, Willett WC, Rimm EB. Prospective study of selenium levels in toenails and risk of coronary heart disease in men. Am J Epidemiol. 2003 Nov 1;158(9):852-60. doi: 10.1093/aje/kwg052. PMID 14585763
- [Background] Koh-Banerjee P, Chu NF, Spiegelman D, Rosner B, Colditz G, Willett W, Rimm E. Prospective study of the association of changes in dietary intake, physical activity, alcohol consumption, and smoking with 9-y gain in waist circumference among 16 587 US men. Am J Clin Nutr. 2003 Oct;78(4):719-27. doi: 10.1093/ajcn/78.4.719. PMID 14522729
- [Background] He K, Merchant A, Rimm EB, Rosner BA, Stampfer MJ, Willett WC, Ascherio A. Dietary fat intake and risk of stroke in male US healthcare professionals: 14 year prospective cohort study. BMJ. 2003 Oct 4;327(7418):777-82. doi: 10.1136/bmj.327.7418.777. PMID 14525873
- [Background] Hung HC, Willett W, Ascherio A, Rosner BA, Rimm E, Joshipura KJ. Tooth loss and dietary intake. J Am Dent Assoc. 2003 Sep;134(9):1185-92. doi: 10.14219/jada.archive.2003.0353. PMID 14528990
- [Background] Hung HC, Merchant A, Willett W, Ascherio A, Rosner BA, Rimm E, Joshipura KJ. The association between fruit and vegetable consumption and peripheral arterial disease. Epidemiology. 2003 Nov;14(6):659-65. doi: 10.1097/01.ede.0000086882.59112.9d. PMID 14569180
- [Background] Newby PK, Hu FB, Rimm EB, Smith-Warner SA, Feskanich D, Sampson L, Willett WC. Reproducibility and validity of the Diet Quality Index Revised as assessed by use of a food-frequency questionnaire. Am J Clin Nutr. 2003 Nov;78(5):941-9. doi: 10.1093/ajcn/78.5.941. PMID 14594780
- [Background] Merchant AT, Pitiphat W, Ahmed B, Kawachi I, Joshipura K. A prospective study of social support, anger expression and risk of periodontitis in men. J Am Dent Assoc. 2003 Dec;134(12):1591-6. doi: 10.14219/jada.archive.2003.0104. PMID 14719755
- [Background] Salazar-Martinez E, Willett WC, Ascherio A, Manson JE, Leitzmann MF, Stampfer MJ, Hu FB. Coffee consumption and risk for type 2 diabetes mellitus. Ann Intern Med. 2004 Jan 6;140(1):1-8. doi: 10.7326/0003-4819-140-1-200401060-00005. PMID 14706966
- [Background] Lopez-Ridaura R, Willett WC, Rimm EB, Liu S, Stampfer MJ, Manson JE, Hu FB. Magnesium intake and risk of type 2 diabetes in men and women. Diabetes Care. 2004 Jan;27(1):134-40. doi: 10.2337/diacare.27.1.134. PMID 14693979
- [Background] He K, Merchant A, Rimm EB, Rosner BA, Stampfer MJ, Willett WC, Ascherio A. Folate, vitamin B6, and B12 intakes in relation to risk of stroke among men. Stroke. 2004 Jan;35(1):169-74. doi: 10.1161/01.STR.0000106762.55994.86. Epub 2003 Dec 11. PMID 14671243
- [Background] Merchant AT, Hu FB, Spiegelman D, Willett WC, Rimm EB, Ascherio A. Dietary fiber reduces peripheral arterial disease risk in men. J Nutr. 2003 Nov;133(11):3658-63. doi: 10.1093/jn/133.11.3658. PMID 14608090
- [Background] Schulze MB, Rimm EB, Shai I, Rifai N, Hu FB. Relationship between adiponectin and glycemic control, blood lipids, and inflammatory markers in men with type 2 diabetes. Diabetes Care. 2004 Jul;27(7):1680-7. doi: 10.2337/diacare.27.7.1680. PMID 15220246
- [Background] Cho E, Seddon JM, Rosner B, Willett WC, Hankinson SE. Prospective study of intake of fruits, vegetables, vitamins, and carotenoids and risk of age-related maculopathy. Arch Ophthalmol. 2004 Jun;122(6):883-92. doi: 10.1001/archopht.122.6.883. PMID 15197064
- [Background] Koh-Banerjee P, Wang Y, Hu FB, Spiegelman D, Willett WC, Rimm EB. Changes in body weight and body fat distribution as risk factors for clinical diabetes in US men. Am J Epidemiol. 2004 Jun 15;159(12):1150-9. doi: 10.1093/aje/kwh167. PMID 15191932
- [Background] Kang JH, Pasquale LR, Willett WC, Rosner BA, Egan KM, Faberowski N, Hankinson SE. Dietary fat consumption and primary open-angle glaucoma. Am J Clin Nutr. 2004 May;79(5):755-64. doi: 10.1093/ajcn/79.5.755. PMID 15113712
- [Background] Choi HK, Atkinson K, Karlson EW, Willett W, Curhan G. Alcohol intake and risk of incident gout in men: a prospective study. Lancet. 2004 Apr 17;363(9417):1277-81. doi: 10.1016/S0140-6736(04)16000-5. PMID 15094272
- [Background] Platz EA, Leitzmann MF, Hollis BW, Willett WC, Giovannucci E. Plasma 1,25-dihydroxy- and 25-hydroxyvitamin D and subsequent risk of prostate cancer. Cancer Causes Control. 2004 Apr;15(3):255-65. doi: 10.1023/B:CACO.0000024245.24880.8a. PMID 15090720
- [Background] Pischon T, Girman CJ, Hotamisligil GS, Rifai N, Hu FB, Rimm EB. Plasma adiponectin levels and risk of myocardial infarction in men. JAMA. 2004 Apr 14;291(14):1730-7. doi: 10.1001/jama.291.14.1730. PMID 15082700
- [Background] Schulze MB, Rimm EB, Li T, Rifai N, Stampfer MJ, Hu FB. C-reactive protein and incident cardiovascular events among men with diabetes. Diabetes Care. 2004 Apr;27(4):889-94. doi: 10.2337/diacare.27.4.889. PMID 15047644
- [Background] Al-Delaimy WK, Rimm EB, Willett WC, Stampfer MJ, Hu FB. Magnesium intake and risk of coronary heart disease among men. J Am Coll Nutr. 2004 Feb;23(1):63-70. doi: 10.1080/07315724.2004.10719344. PMID 14963055
- [Background] Pai JK, Pischon T, Ma J, Manson JE, Hankinson SE, Joshipura K, Curhan GC, Rifai N, Cannuscio CC, Stampfer MJ, Rimm EB. Inflammatory markers and the risk of coronary heart disease in men and women. N Engl J Med. 2004 Dec 16;351(25):2599-610. doi: 10.1056/NEJMoa040967. PMID 15602020
- [Background] Bohler J, Woitas R, Keller E, Reetze-Bonorden P, Schollmeyer PJ. Effect of nifedipine and captopril on glomerular hyperfiltration in normotensive man. Am J Kidney Dis. 1992 Aug;20(2):132-9. doi: 10.1016/s0272-6386(12)80540-3. PMID 1496965
- [Background] Mozaffarian D, Ascherio A, Hu FB, Stampfer MJ, Willett WC, Siscovick DS, Rimm EB. Interplay between different polyunsaturated fatty acids and risk of coronary heart disease in men. Circulation. 2005 Jan 18;111(2):157-64. doi: 10.1161/01.CIR.0000152099.87287.83. Epub 2005 Jan 3. PMID 15630029
- [Background] Mukamal KJ, Ascherio A, Mittleman MA, Conigrave KM, Camargo CA Jr, Kawachi I, Stampfer MJ, Willett WC, Rimm EB. Alcohol and risk for ischemic stroke in men: the role of drinking patterns and usual beverage. Ann Intern Med. 2005 Jan 4;142(1):11-9. doi: 10.7326/0003-4819-142-1-200501040-00007. PMID 15630105
- [Background] Eng PM, Kawachi I, Fitzmaurice G, Rimm EB. Effects of marital transitions on changes in dietary and other health behaviours in US male health professionals. J Epidemiol Community Health. 2005 Jan;59(1):56-62. doi: 10.1136/jech.2004.020073. PMID 15598728
- [Background] Jensen MK, Koh-Banerjee P, Hu FB, Franz M, Sampson L, Gronbaek M, Rimm EB. Intakes of whole grains, bran, and germ and the risk of coronary heart disease in men. Am J Clin Nutr. 2004 Dec;80(6):1492-9. doi: 10.1093/ajcn/80.6.1492. PMID 15585760
- [Background] Pitiphat W, Crohin C, Williams P, Merchant AT, Douglass CW, Colditz GA, Joshipura KJ. Use of preexisting radiographs for assessing periodontal disease in epidemiologic studies. J Public Health Dent. 2004 Fall;64(4):223-30. doi: 10.1111/j.1752-7325.2004.tb02757.x. PMID 15562945
- [Background] Hung HC, Joshipura KJ, Colditz G, Manson JE, Rimm EB, Speizer FE, Willett WC. The association between tooth loss and coronary heart disease in men and women. J Public Health Dent. 2004 Fall;64(4):209-15. doi: 10.1111/j.1752-7325.2004.tb02755.x. PMID 15562943
- [Background] Koh-Banerjee P, Franz M, Sampson L, Liu S, Jacobs DR Jr, Spiegelman D, Willett W, Rimm E. Changes in whole-grain, bran, and cereal fiber consumption in relation to 8-y weight gain among men. Am J Clin Nutr. 2004 Nov;80(5):1237-45. doi: 10.1093/ajcn/80.5.1237. PMID 15531671
- [Background] Hung HC, Joshipura KJ, Jiang R, Hu FB, Hunter D, Smith-Warner SA, Colditz GA, Rosner B, Spiegelman D, Willett WC. Fruit and vegetable intake and risk of major chronic disease. J Natl Cancer Inst. 2004 Nov 3;96(21):1577-84. doi: 10.1093/jnci/djh296. PMID 15523086
- [Background] Shai I, Rimm EB, Schulze MB, Rifai N, Stampfer MJ, Hu FB. Moderate alcohol intake and markers of inflammation and endothelial dysfunction among diabetic men. Diabetologia. 2004 Oct;47(10):1760-7. doi: 10.1007/s00125-004-1526-0. Epub 2004 Oct 22. PMID 15502925
- [Background] Rajpathak S, Rimm EB, Li T, Morris JS, Stampfer MJ, Willett WC, Hu FB. Lower toenail chromium in men with diabetes and cardiovascular disease compared with healthy men. Diabetes Care. 2004 Sep;27(9):2211-6. doi: 10.2337/diacare.27.9.2211. PMID 15333486
- [Background] Jiang R, Schulze MB, Li T, Rifai N, Stampfer MJ, Rimm EB, Hu FB. Non-HDL cholesterol and apolipoprotein B predict cardiovascular disease events among men with type 2 diabetes. Diabetes Care. 2004 Aug;27(8):1991-7. doi: 10.2337/diacare.27.8.1991. PMID 15277429
- [Background] Al-Delaimy WK, Merchant AT, Rimm EB, Willett WC, Stampfer MJ, Hu FB. Effect of type 2 diabetes and its duration on the risk of peripheral arterial disease among men. Am J Med. 2004 Feb 15;116(4):236-40. doi: 10.1016/j.amjmed.2003.09.038. PMID 14969651
- [Background] Joshipura KJ, Wand HC, Merchant AT, Rimm EB. Periodontal disease and biomarkers related to cardiovascular disease. J Dent Res. 2004 Feb;83(2):151-5. doi: 10.1177/154405910408300213. PMID 14742654
- [Background] Kang JH, Pasquale LR, Rosner BA, Willett WC, Egan KM, Faberowski N, Hankinson SE. Prospective study of cigarette smoking and the risk of primary open-angle glaucoma. Arch Ophthalmol. 2003 Dec;121(12):1762-8. doi: 10.1001/archopht.121.12.1762. PMID 14662597
- [Background] Wang Y, Rimm EB, Stampfer MJ, Willett WC, Hu FB. Comparison of abdominal adiposity and overall obesity in predicting risk of type 2 diabetes among men. Am J Clin Nutr. 2005 Mar;81(3):555-63. doi: 10.1093/ajcn/81.3.555. PMID 15755822
- [Background] Choi HK, Willett WC, Stampfer MJ, Rimm E, Hu FB. Dairy consumption and risk of type 2 diabetes mellitus in men: a prospective study. Arch Intern Med. 2005 May 9;165(9):997-1003. doi: 10.1001/archinte.165.9.997. PMID 15883237
- [Background] Qi L, Rimm E, Liu S, Rifai N, Hu FB. Dietary glycemic index, glycemic load, cereal fiber, and plasma adiponectin concentration in diabetic men. Diabetes Care. 2005 May;28(5):1022-8. doi: 10.2337/diacare.28.5.1022. PMID 15855561
- [Background] Qi L, Li T, Rimm E, Zhang C, Rifai N, Hunter D, Doria A, Hu FB. The +276 polymorphism of the APM1 gene, plasma adiponectin concentration, and cardiovascular risk in diabetic men. Diabetes. 2005 May;54(5):1607-10. doi: 10.2337/diabetes.54.5.1607. PMID 15855354
- [Background] Hung HC, Colditz G, Joshipura KJ. The association between tooth loss and the self-reported intake of selected CVD-related nutrients and foods among US women. Community Dent Oral Epidemiol. 2005 Jun;33(3):167-73. doi: 10.1111/j.1600-0528.2005.00200.x. PMID 15853839
- [Background] Pischon T, Girman CJ, Rifai N, Hotamisligil GS, Rimm EB. Association between dietary factors and plasma adiponectin concentrations in men. Am J Clin Nutr. 2005 Apr;81(4):780-6. doi: 10.1093/ajcn/81.4.780. PMID 15817852
- [Background] Schulze MB, Shai I, Rimm EB, Li T, Rifai N, Hu FB. Adiponectin and future coronary heart disease events among men with type 2 diabetes. Diabetes. 2005 Feb;54(2):534-9. doi: 10.2337/diabetes.54.2.534. PMID 15677512
- [Background] Mukamal KJ, Jensen MK, Gronbaek M, Stampfer MJ, Manson JE, Pischon T, Rimm EB. Drinking frequency, mediating biomarkers, and risk of myocardial infarction in women and men. Circulation. 2005 Sep 6;112(10):1406-13. doi: 10.1161/CIRCULATIONAHA.105.537704. Epub 2005 Aug 29. PMID 16129796
- [Background] Pischon T, Girman CJ, Sacks FM, Rifai N, Stampfer MJ, Rimm EB. Non-high-density lipoprotein cholesterol and apolipoprotein B in the prediction of coronary heart disease in men. Circulation. 2005 Nov 29;112(22):3375-83. doi: 10.1161/CIRCULATIONAHA.104.532499. PMID 16316964
- [Background] Giovannucci E, Willett WC. Dietary factors and risk of colon cancer. Ann Med. 1994 Dec;26(6):443-52. doi: 10.3109/07853899409148367. PMID 7695871
- [Background] Hemenway D, Azrael DR, Rimm EB, Feskanich D, Willett WC. Risk factors for hip fracture in US men aged 40 through 75 years. Am J Public Health. 1994 Nov;84(11):1843-5. doi: 10.2105/ajph.84.11.1843. PMID 7977932
- [Background] Giovannucci E, Rimm EB, Stampfer MJ, Colditz GA, Willett WC. Height, body weight, and risk of prostate cancer. Cancer Epidemiol Biomarkers Prev. 1997 Aug;6(8):557-63. PMID 9264267
- [Background] Hu FB, Stampfer MJ, Rimm EB, Manson JE, Ascherio A, Colditz GA, Rosner BA, Spiegelman D, Speizer FE, Sacks FM, Hennekens CH, Willett WC. A prospective study of egg consumption and risk of cardiovascular disease in men and women. JAMA. 1999 Apr 21;281(15):1387-94. doi: 10.1001/jama.281.15.1387. PMID 10217054
- [Derived] Liu X, Guasch-Ferre M, Drouin-Chartier JP, Tobias DK, Bhupathiraju SN, Rexrode KM, Willett WC, Sun Q, Li Y. Changes in Nut Consumption and Subsequent Cardiovascular Disease Risk Among US Men and Women: 3 Large Prospective Cohort Studies. J Am Heart Assoc. 2020 Apr 7;9(7):e013877. doi: 10.1161/JAHA.119.013877. Epub 2020 Apr 1. PMID 32233756
- [Derived] Zong G, Liu G, Willett WC, Wanders AJ, Alssema M, Zock PL, Hu FB, Sun Q. Associations Between Linoleic Acid Intake and Incident Type 2 Diabetes Among U.S. Men and Women. Diabetes Care. 2019 Aug;42(8):1406-1413. doi: 10.2337/dc19-0412. Epub 2019 Jun 10. PMID 31182488
- [Derived] Liu X, Li Y, Tobias DK, Wang DD, Manson JE, Willett WC, Hu FB. Changes in Types of Dietary Fats Influence Long-term Weight Change in US Women and Men. J Nutr. 2018 Nov 1;148(11):1821-1829. doi: 10.1093/jn/nxy183. PMID 30247611
- [Derived] Zong G, Li Y, Sampson L, Dougherty LW, Willett WC, Wanders AJ, Alssema M, Zock PL, Hu FB, Sun Q. Monounsaturated fats from plant and animal sources in relation to risk of coronary heart disease among US men and women. Am J Clin Nutr. 2018 Mar 1;107(3):445-453. doi: 10.1093/ajcn/nqx004. PMID 29566185